CLINICAL TRIAL: NCT06375642
Title: A Single Arm, Single Centered Phase II Trial on the Combination of Adebrelimab, Surufatinib and Irinotecan Liposome-based Hepatic Artery Infusion Chemotherapy in the Treatment of Advanced Intrahepatic Cholangiocarcinoma
Brief Title: A Single Arm, Single Centered Phase II Trial on the Combination of Adebrelimab, Surufatinib and Irinotecan Liposome-based HAIC in Advanced iCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, HuiKai Li, Chief Physician, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR1316-HMPL012-HAIC-01
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Surufatinib: 100 mg orally qd, Adebrelimab: 1200 mg, IV, q3w, HAIC: Irinotecan liposome 30 mg/m2, leucovorin 200 mg/m2, 5-FU 200 mg/m2 bolus followed by continuous infusion of 5-FU 1200 mg/m2 5-FU q3W for 24 h. Dose adjustment was allowed for instilled drugs during treatment, and delayed administration was allowed for up to 8 weeks, calculated from the last administration time, otherwise treatment was terminated.
  Tumor assessment will be performed by imaging method every 3 cycles (± 7 days) in 21-day cycles until disease progression (RECIST 1.1) or death (during treatment), and tumor treatment and survival status after disease progression will be recorded.
  Interventions: Drug: Adebrelimab

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab, Surufatinib and HAIC
  Other Names: Surufatinib; HAIC

SUMMARY:
Southeast Asia and China have the highest incidence of intrahepatic cholangiocarcinoma worldwide, with limited treatment options and large unmet medical needs.

Hepatic arterial infusion chemotherapy (HAIC) has gradually emerged as a promising treatment option for patients with hepatocellular carcinoma (HCC). Increasing evidence suggests that infusion of HAIC, which maintains high local concentrations of toxic agents in tumors without embolism, provides a significant survival benefit for patients with advanced HCC and is well-tolerated. However, there is limited evidence for the efficacy of HAIC for intrahepatic cholangiocarcinoma.

Irinotecan liposome (nal-IRI) is a concentrate of an infusion solution containing 5 mg/ml irinotecan trihydrate (irinotecan sucrose salt) active substance, which is encapsulated in liposomes and prevents premature conversion of the drug to SN-38 in the liver. Liposomal irinotecan prolongs the circulation time of the drug in the plasma of patients and prolongs the tumor exposure of the drug compared to conventional irinotecan.Nal-IRI based protocol has shown positive results in the phase III trial of pancreatic carcinoma.

Adebrelima(SHR-1316) is a recombinant humanized IgG4 antibody that binds efficiently and specifically to human and cynomolgus programmed cell death ligand 1 (PD-L1, CD274, or B7-H1), a cell surface molecule that plays an important role in T cell immune function, and stimulates IFN-γ secretion from mixed lymphocyte reactions (MLRs) of dendritic cells (DCs) and CD4 + T cells.

Surufatinib is a multiple kinase inhibitor targeting VEGFR 1-3, FGFR1 and CSF1R.

This study aims to evaluate the efficacy and safety of irinotecan liposome-based hepatic arterial infusion chemotherapy combined with adebrelimab and surufatinib in the treatment of intrahepatic cholangiocarcinoma, which may bring significant clinical benefit to the iCC patients with new treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form before enrollment;
2. Age > 18 years, both men and women;
3. Patients with histologically or pathologically confirmed intrahepatic cholangiocarcinoma;
4. No previous systemic therapy and local therapy;
5. Measurable intrahepatic lesions (according to RECIST 1.1 criteria, the long diameter of CT scan of non-lymph node lesions is ≥ 10 mm, and the short diameter of CT scan of lymph node lesions is ≥ 15 mm);
6. ECOG PS score: 0-1;
7. Expected survival greater than 12 weeks;
8. Vital organs function in accordance with the following requirements (excluding any blood components and cell growth factors used within 14 days):

1) Blood routine: Neutrophils ≥ 1.5 × 109/L; Platelet count ≥ 60 × 109/L;Hemoglobin ≥ 90 g/L; 2) Hepatic and renal function: Serum creatinine (SCr) ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula);Total bilirubin (TBIL) ≤ 3 times the upper limit of normal (ULN);Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤ 10 times the upper limit of normal (ULN); urine protein < 2 +; if urine protein ≥ 2 +, 24-hour urine protein quantification must show protein ≤ 1 g; 9. Normal coagulation function, no active bleeding and thrombosis disease

1. International normalized ratio INR ≤ 1.5 × ULN;
2. Partial thromboplastin time APTT ≤ 1.5 × ULN;
3. PT ≤ 1.5 × ULN; 10. Non-surgically sterilized or female patients of childbearing age need to use a medically recognized contraceptive (such as intrauterine device, contraceptives or condoms) during study treatment and within 3 months after the end of study treatment; non-surgically sterilized female patients of childbearing age must have a negative serum or urine HCG test within 7 days before study enrollment; and must be non-lactating; non-surgically sterilized or male patients of childbearing age need to agree to use a medically recognized contraceptive during study treatment and within 3 months after the end of study treatment with their spouses.

11. The subject voluntarily joins this study, has good compliance, and cooperates with safety and survival follow-up

Exclusion Criteria:

1. The subject has previous or concurrent other malignancies (except cured cutaneous basal cell carcinoma and cervical carcinoma in situ);
2. Previous immunotherapy except anti-PD-1/PD-L1 monoclonal antibody; known subject has previously been allergic to macromolecular protein preparations, or known hypersensitivity to the applied drug components;
3. Subjects with any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, previous thyroid surgery can not be included; subjects with vitiligo or childhood asthma has been completely relieved, no intervention is required after adults can be included; subjects with asthma requiring bronchodilators for medical intervention can not be included);
4. Subjects are using immunosuppressive agents, or systemic, or absorbable local hormone therapy to achieve immunosuppressive purposes (dose > 10 mg/day prednisone or other effective hormones), and continue to use within 2 weeks before enrollment;
5. Ascites or pleural effusion with clinical symptoms, ascites requiring therapeutic puncture or regular drainage (≥ 1 time/month);
6. Patients with poorly controlled cardiac clinical symptoms or diseases, such as: (1) NYHA2 or higher heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
7. The subject has active infection or unexplained fever > 38.5 degrees during screening or before the first dose (the subject can be enrolled due to fever caused by the tumor as judged by the investigator);
8. Patients with previous and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired pulmonary function;
9. Subjects with congenital or acquired immunodeficiency, such as HIV infection;
10. Live vaccines less than 4 weeks before study drug or likely during the study;
11. The subject has a known history of psychiatric drug abuse, alcoholism or drug abuse;
12. Patients who cannot be orally administered;
13. Received Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 2 weeks before the first dose.
14. The investigator believes that the subject should be excluded from this study, for example, the investigator judges that the subject has other factors that may cause forced halfway termination of this study, for example, other serious diseases (including mental illness) require concomitant treatment, severe gastroesophageal varices, serious laboratory abnormalities, accompanied by family or social factors, which may affect the safety of the subject, or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From treatment initiation to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease(PD), using RECIST v1.1
Disease Control Rate | From treatment initiation to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease(PD), using RECIST v1.1

SECONDARY OUTCOMES:
Overall Survival | from treatment initiation until death due to any cause, assessed up to 3 year
  every two months follow up after EOT observation period at 30 days after the last medication
Progress-Free Survival | from treatment initiation until death due to any cause, assessed up to 2 year
  every two months follow up after EOT observation period at 30 days after the last medication
Incidence and severity of AE and SAE | from first dose to 30 days post the last dose
  Safety
Dose suspension rate caused by adverse events | from first dose to 30 days post the last dose
  Safety
dose termination rate caused by adverse events | from first dose to 30 days post the last dose
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No